CLINICAL TRIAL: NCT04487496
Title: Determinants of Access to Emergency Surgery at the University College Hospital, Ibadan
Status: Completed | Type: Observational
Sponsor: University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, Dr. Promise Tamunoipiriala Jaja, Doctor, University College Hospital, Ibadan
Other Study IDs: U1111-1254-0480
Record Dates: First submitted 2020-06-22; First posted 2020-07-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Access to Emergency Surgery
Keywords: Emergency surgery; Access to emergency surgery; Acute surgical care; Acute trauma care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Access to surgery is reported to be significantly lower in low income countries like Nigeria, and upwards of 5 billion people globally lack safe access to surgery. The investigators intend to answer the question, what is the burden of access to acute care surgery alongside their determinants in the University College Hospital, Ibadan (UCH). The expected results from this study will provide basis for evidence-based policy aimed at improving time-to-emergency surgery and thus improve outcomes.

A cross-sectional doctors' survey and a prospective case records review would be the study designs; using a minimum of fifty-one participants and case records respectively. The doctors will be selected randomly from all the surgical services and the emergency department in the UCH, ensuring a fairly equal allocation. The case notes will be of patients in the UCH requiring emergency surgery that had surgeries.

Data from this study will be entered and analysed using STATA/MP 15.0 (Stata Corp, College station, TX).

DETAILED DESCRIPTION:
Introduction The Sustainable Development Goals (SDG) mandates that to improve health and health equity, every global citizen has a right to improved essential and emergency surgical care and States are morally obliged to ensure this (Chawla, Rutkov, Garber, Kushner, & Stewart, 2017). These were ratified by the World Health Assembly Resolution 68.15 that made access to quality and timely Emergency and Essential Surgical Care and Anaesthesia (EESCA) a component of the Universal Health Coverage (Chawla, Rutkov, Garber, Kushner, & Stewart, 2017). It is accepted that prompt access to surgical care is cardinal for the reduction of the potentially associated morbidity and mortality inherent in surgical conditions (Scott, et al., 2016). Care following trauma has been proposed as a model for accessing indiscriminate care, as care seeking here is mostly guided by injury severity (Scott, et al., 2016); hence, we would use trauma related metrics to present a rationale for this study.

Civilian trauma mortality have been postulated to follow the so-called tri-modal death peaks, 50% of those mortalities -representing the first peak- present emergency care physicians with the dilemma of almost sudden death (occurring within seconds to minutes), thus they very rarely survive past the trauma field (Solomon, Warwick, & Nayagam, 2010). The other 50% is distributed as 30% and 20% for the second and third peaks respectively. These casualties are actually capable of presenting for care, as the second peak deaths will occur within minutes to hours and is nicknamed 'Golden hour' because a carefully executed trauma algorithm will ensure to avert a mortality in that situation; attention here is placed on carefully identifying potentially catastrophic haemorrhage of the overt or covert forms, the efficient and rapid establishment of haemostasis and treatment of circulatory shock (Solomon, Warwick, & Nayagam, 2010). The third peak deaths may represent a failure of preventing and treating infections as well as failure to co-manage other morbidities in these patients; there is a resultant two-week interval before such septic processes are significantly established to threaten survival of the post-acute phase trauma patient (World health statistics 2019: monitoring health for the SDGs, sustainable development goals. Licence: CC BY-NC-SA 3.0 IGO., 2019; Solomon, Warwick, & Nayagam, 2010).

Statement of problem Poisoning, motor vehicle crashes and firearm injuries are the leading causes of Emergency Room (ER) visits in the United States of America (USA); clearly, with the exception of poisoning, trauma-related causes necessitate most visits in the USA, in accordance with reports of trauma being the leading cause of death for persons under 45 years of age in the USA (Gani, Sakran, & Canner, 2017; Carr, et al., 2017). The annual trauma-related ER visits in the US are about 29 million visits, resulting in 2.8 million hospitalizations and 180 thousand deaths (Carr, et al., 2017) and the American region's Road Traffic Mortality Rate (RTMR) at 15.6 per 100,000 (World health statistics 2019: monitoring health for the SDGs, sustainable development goals. Licence: CC BY-NC-SA 3.0 IGO., 2019). These are despite that 88.3% of the American population have access to high level trauma centres (Carr, et al., 2017), the American region has a Universal Health Coverage (UHC) service coverage index of 78% and Density of Medical Doctors (DMD) of 23.3 per 10,000 population.

It is worthy of note that globally, five billion people lack access to safe and affordable surgery when needed, irrespective of the fact that globally 312 million surgical procedures are done annually, only about 6% of these are done in the poorest countries (Watters, Guest, Tangi, Shrime, & Meara, 2018). This is against the fact that in 2016 the low and middle income earning countries account for 93% of the 1.3 million people reported to have had road traffic accidents (RTA) and the upwards of 50 million people that were injured (World health statistics 2019: monitoring health for the SDGs, sustainable development goals. Licence: CC BY-NC-SA 3.0 IGO., 2019). Their survival may have been improved if the Healthy people 2020 benchmark on access to trauma care of 60 minutes could be met (Carr, et al., 2017); well this isn't the case as in 2016, RTMR per 100,000 population was 26.6, 27.5 and 19.2 in the African region, low and middle income earning countries unlike 8.3 in the high income earning countries and the UHC service coverage indices were 44%, 78% and 73% respectively for the African, American and European regions respectively and a similar tale for the DMD per 10,000 population at 2.8, 23.3 and 33.8 for the African, American and European regions respectively (World health statistics 2019: monitoring health for the SDGs, sustainable development goals. Licence: CC BY-NC-SA 3.0 IGO., 2019).

Aim of the study The study aims to identify the determinants of access to emergency surgeries in the University College Hospital Ibadan

Objectives of the study

General: To establish the determinants of access to emergency surgeries at the University College Hospital Ibadan

Specific:

To establish the average time-to-surgery for surgical emergencies in the University College Hospital Ibadan To establish the burden of delayed emergency surgeries in University College Hospital Ibadan.

To determine the patient related causes of delayed emergency surgeries in the University College Hospital Ibadan.

To elucidate the healthcare giver related causes of delayed emergency surgeries in the University College Hospital Ibadan.

To examine the institutional factors related to the causes of delayed emergency surgeries in the University College Hospital Ibadan.

To aggregate the determinants of causes of delayed emergency surgeries in the University College Hospital Ibadan and present a multivariate analysis of their inter-relation.

ELIGIBILITY:
Inclusion Criteria:

* All recruited doctors who give consent
* All eligible case records of surgical emergencies determined by the surgical services.

Exclusion Criteria:

* Case records of patients to be directly managed by the principal investigator
* Case records of patients who die before surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This shall comprise all the healthcare givers related to the surgical specialties in UCH, these include the following departments: surgery, plastics and reconstructive and aesthetic surgery, neurological surgery, orthopaedics and trauma, otorhinolaryngology, ophthalmology, obstetrics and gynaecology, oral and maxillofacial surgery, anaesthesia as well as the accident and emergency.
  The case-records of all patients presenting through the emergency room of University College Hospital Ibadan, requiring emergency surgery as determined by the surgical services.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Time-to-surgery | One year
  This will collect information about the time from specific event (onset of symptoms, entry into the hospital, diagnosis and decision for surgical care) to the actual onset of the emergency surgery
Factors affecting onset of emergency surgery | One year
  This will gather from the doctors' survey and the prospective case records review, the patient related, healthcare giver related and institutional related determinants of access to emergency surgery

SECONDARY OUTCOMES:
Post-operative outcome | One year
  This will collect outcome data from the case records review, these will include the presence or absence of post-operative complications, the length of hospital stay and final disposition of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Promise T Jaja, MB;BS, MSc, Principal Investigator — University College Hospital, Ibadan; Adefemi O Afolabi, MB;BS, FWACS, Study Director — University College Hospital, Ibadan
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set will be developed and presented in a share-able format and most likely deposited in an online data repository
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available within two years of the final completion of the study
Access Criteria: Access will be granted following a review of written requests for the data

REFERENCES:
- [Background] Carr BG, Bowman AJ, Wolff CS, Mullen MT, Holena DN, Branas CC, Wiebe DJ. Disparities in access to trauma care in the United States: A population-based analysis. Injury. 2017 Feb;48(2):332-338. doi: 10.1016/j.injury.2017.01.008. Epub 2017 Jan 3. PMID 28069138
- [Background] Chawla KS, Rutkow L, Garber K, Kushner AL, Stewart BT. Beyond a Moral Obligation: A Legal Framework for Emergency and Essential Surgical Care and Anesthesia. World J Surg. 2017 May;41(5):1208-1217. doi: 10.1007/s00268-016-3866-6. PMID 28180984
- [Background] Gani F, Sakran JV, Canner JK. Emergency Department Visits For Firearm-Related Injuries In The United States, 2006-14. Health Aff (Millwood). 2017 Oct 1;36(10):1729-1738. doi: 10.1377/hlthaff.2017.0625. PMID 28971917
- [Background] MC, R. (1991). An in-vivo of the microbial proliferation beneath transport film dressings in: Maki DG, ed, International congress and symposium series No 179, improving catheter site care. London Series (pp. 29-33). London: Royal Society of Medicine.
- [Background] Scott JW, Havens JM, Wolf LL, Zogg CK, Rose JA, Salim A, Haider AH. Insurance status is associated with complex presentation among emergency general surgery patients. Surgery. 2017 Feb;161(2):320-328. doi: 10.1016/j.surg.2016.08.038. Epub 2016 Oct 4. PMID 27712875
- [Background] Solomon, L., Warwick, D., & Nayagam, S. (2010). Apley's System of Orthopaedics and Fractures. London: Hodder Arnold.
- [Background] Watters DA, Guest GD, Tangi V, Shrime MG, Meara JG. Global Surgery System Strengthening: It Is All About the Right Metrics. Anesth Analg. 2018 Apr;126(4):1329-1339. doi: 10.1213/ANE.0000000000002771. PMID 29547428
- [Background] World health statistics 2019: monitoring health for the SDGs, sustainable development goals. Licence: CC BY-NC-SA 3.0 IGO. (2019). Geneva: World Health Organization. Retrieved August 15, 2019, from https://www.who.int/gho/publications/world_health_statistics/2019/EN_WHS_2019_Main.pdf?ua=1